CLINICAL TRIAL: NCT05540262
Title: Edaravone in the Treatment of Optic Neuritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yi Du, Dr., First Affiliated Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GXEDAON1.0
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis | interventions — Edaravone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Edaravone (Experimental)
  Interventions: Drug: Edaravone

INTERVENTIONS:
Drug: Edaravone — Edaravone injection 30mg three times a day

SUMMARY:
Edaravone has demonstrated a beneficial effect in promoting remyelination and protecting axons in animals with NMOSD. The researchers posit that edaravone may enhance visual outcomes in patients with aquaporin-4 antibody-positive optic neuritis.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese patients aged ≥18 with anti-aquaporin-4 antibody-positive optic neuritis
2. Patients with a first episode of optic neuritis in either eye
3. First symptoms of optic neuritis ≤30 days prior to the first administration of edaravone

Exclusion Criteria:

1. Myopia over 6 diopters
2. Refractive media opacity affecting assessment of retinal layers and/or visual acuity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity | 18 months
  Best-corrected visual acuity will be measured by "Illiterate E"chart.

SECONDARY OUTCOMES:
Ganglion cell-inner plexiform layer | 18 months
  Ganglion cell-inner plexiform layer will be measured by optical coherence tomography.
Peripapillary retinal nerve fiber layer | 18 months
  Peripapillary retinal nerve fiber layer will be measured by optical coherence tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- Yi Du, Nanning, China

IPD SHARING:
Plan to Share IPD: Undecided